CLINICAL TRIAL: NCT05700201
Title: The Effects of a Cognitive Behavioral Healthy Lifestyle Intervention for Cardiovascular Risk Reduction in Posttraumatic Stress Disorder
Brief Title: Investigating Cardiac Health of Adults With Trauma
Acronym: I - CHAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Jeffrey Kibler, Ph.D., Professor, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R15HL165308-01 (NIH)
Record Dates: First submitted 2023-01-04; First posted 2023-01-26 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress; Cardiovascular; Health; Intervention; PTSD; Lifestyle; Behavior
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Behavior | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study involves examining the effects of a 12-session healthy lifestyle program (focused on physical activity, nutrition, sleep, and stress management) administered in an individual format as an adjunct to usual care psychotherapy, compared with a usual care psychotherapy-only control condition. The control group will only attend the outcome assessments and usual care psychotherapy sessions. Therefore, the design relies on a between-groups comparison of the two conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Healthy lifestyle intervention
  Interventions: Behavioral: Lifestyle / Healthy Behavior Intervention
- Control (Experimental): Standard care (psychotherapy)
  Interventions: Other: standard care

INTERVENTIONS:
Behavioral: Lifestyle / Healthy Behavior Intervention — 12-session healthy lifestyle program focused on physical activity, nutrition, sleep, and stress management.
  Arms: Intervention
Other: standard care — Standard care (psychotherapy)
  Arms: Control

SUMMARY:
This project examines the impact of a healthy lifestyle intervention, specifically designed for adults with posttraumatic stress and identified cardiovascular risks.

DETAILED DESCRIPTION:
Considerable research has indicated strong associations between posttraumatic stress and cardiovascular disease (CVD) risk. Individuals with posttraumatic stress disorder (PTSD) tend to show patterns of elevated CVD risk earlier in life than in the general population. The need for developing effective interventions for CVD risk-reduction in PTSD is increasingly evident. In comparison to the cumulative evidence concerning elevated CVD risk in PTSD, relatively little research has addressed CVD risk-reduction in this population. Adjunctive treatments, such as health behavior interventions, may be necessary as supplements to traditional psychotherapy for PTSD in order to reduce CVD risks. The objective of the proposed project is to examine the effects of a healthy lifestyle intervention that addresses multiple CVD-related heath behaviors among civilian adults across genders (ages 18+), who evidence PTSD and CVD risk at baseline. The investigators will assess the intervention impact on both subjective and objective indices of health behaviors, cardiovascular risks and CVD markers over a one-year timeframe. The healthy lifestyle intervention addresses unique aspects of PTSD symptom presentation that serve as barriers to healthy behaviors (e.g., nightmares/sleep disruption, and cognitive responses to stress), while encouraging healthy lifestyle changes. The primary goal of the present study is to examine whether, compared to a usual care psychotherapy control condition, utilizing the healthy lifestyle intervention as an adjunct to psychotherapy will result in significantly reduced CVD risks and improved CVD markers among civilian adults with PTSD and elevated CVD risks. Therefore, participants will be randomly assigned to either a usual care psychotherapy-only control condition or a usual care psychotherapy plus healthy lifestyle intervention condition. Outcomes will be assessed at post-intervention (12 weeks), as well as 6-month and 12-month time points for follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* PTSD symptoms
* overweight OR less than 30 min. of moderate physical activity 5 times per week

Exclusion Criteria:

* cannot exercise at a low-moderate level (walking)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 1 year
  The International Physical Activity Questionnaire (7-Day long form) is a reliable and valid measure that will be used to assess time spent in a variety of moderate and vigorous activities in the past week

SECONDARY OUTCOMES:
Arterial Stiffness | 1 year
  non-invasive measurement of augmentation index, calculated as the difference between the second and the first systolic peaks and expressed as percentage of the central aortic pulse pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kibler, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- College of Psychology, Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided